CLINICAL TRIAL: NCT02163876
Title: A Single-Blind, Randomized, Parallel Arm, Phase II Proof-of-Concept Study of the Safety and Efficacy of Human Central Nervous System Stem Cells (HuCNS-SC) Transplantation in Cervical Spinal Cord Injury
Brief Title: Study of Human Central Nervous System (CNS) Stem Cell Transplantation in Cervical Spinal Cord Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on a business decision unrelated to any safety concerns.
Sponsor: StemCells, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL-SCI-201
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Cervical Spinal Cord Injury; Spine Injury; Cervical Spine Injury
Keywords: spine; injury; trauma; spine injury; cervical spine injury; cervical spine; stemcells transplantation
MeSH Terms: conditions — Spinal Injuries; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HuCNS-SC cells (Experimental): Intramedullary transplantation of HuCNS-SC cells in the cervical spine
  Interventions: Drug: HuCNS-SC cells
- non-surgery arm (No Intervention): non-surgery arm

INTERVENTIONS:
Drug: HuCNS-SC cells — surgery arm
  Other Names: human neural stem cells; HuCNS-SC; HCNS-SC
  Arms: HuCNS-SC cells

SUMMARY:
This study will evaluate the safety and efficacy of human central nervous system stem cell transplantation into patients with traumatic injury in the cervical region of the spinal cord.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 18 to 60 years.
* Traumatic cervical spinal cord injury (cSCI) with C5-C7 motor levels according to the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) as determined by the Investigator.
* American Spinal Injury Association Impairment Scale (AIS) Grades B or C
* Minimum of 12 weeks post-injury prior to Screening

Exclusion Criteria:

* History of penetrating SCI.
* MRI evidence of complete spinal cord interruption .
* Evidence of spinal instability, stenosis and/or persistent cord compression related to the initial trauma.
* Prior participation in another investigational study within 90 days prior to Screening.
* Previous organ, tissue, bone marrow transplantation, or gene transfer
* History of malignancy (except non-melanoma skin cancers) that require(d) radiation and/or chemotherapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ISNCSCI upper extremity motor scores | Up to one year after enrollment

SECONDARY OUTCOMES:
Number of participants with serious and non-serious adverse events | Up to one year from the time of enrollment
  Safety measures will include collection of adverse events, laboratory tests, neurological examination, ISNCSCI motor and sensory scores, pain and allodynia assessment, AIS grade, physical examination and modified Ashworth scale

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, MD, Study Director — StemCells, Inc.
Locations (14):
- United States (12):
  - Rancho Los Amigos National Rehabilitation Center/USC, Downey, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Maryland Medical Systems, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota/Courage Kenny Rehabilitation Institute, Minneapolis, Minnesota
  - Mount Sinai Medical Center, Dept of Neurosurgery, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas, Mischer Neuroscience Institute, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Canada (2):
  - Foothills Medical Center, Calgary, Alberta
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Ahuja CS, Fehlings M. Concise Review: Bridging the Gap: Novel Neuroregenerative and Neuroprotective Strategies in Spinal Cord Injury. Stem Cells Transl Med. 2016 Jul;5(7):914-24. doi: 10.5966/sctm.2015-0381. Epub 2016 Apr 29. PMID 27130222
- See also: Spinal Cord Injury Program — http://www.stemcellsinc.com/therapeutic-programs/spinal-cord-injury.htm
- See also: Study Website — https://sciresearchstudy.com